CLINICAL TRIAL: NCT04021732
Title: Effects of Exercise on Metabolic Parameters in Treated Patients With Classical Homocystinuria: a Research Project on a Small Sample Size, Compared to Healthy Controls.
Brief Title: Effects of Exercise on Metabolic Parameters in Classical Homocystinuria
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Christel Tran, Associate physician, University of Lausanne
Other Study IDs: 2018-02400
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-02

CONDITIONS: Homocystinuria
MeSH Terms: conditions — Homocystinuria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this research project is to compare the effect of an aerobic exercise session in two different populations. Sampling biological material and collecting health-related personal data entails minimal risks and burdens. Participants will be asked to perform 30 minutes of an aerobic exercise on an ergocycle at a fixed power output to correspond to a moderate intensity for a sedentary population.

DETAILED DESCRIPTION:
Background Among genetic causes of hyperhomocysteinemia, classical homocystinuria, manifest not only with vascular diseases but also with neurological symptoms. This is related to the higher homocysteine concentration of up to 150-300 μmol/l without treatment. Recently, some articles have shown that mild and temporary hyperhomocysteinemia may follow exercise in a healthy population. Investigators hypothesized that increase in homocysteine may be of greater importance in patients with classical homocystinuria where cystathionine beta-synthase deficiency prevents homocysteine metabolism.

Objective To investigate the effect of an aerobic exercise in patients with classical homocystinuria on metabolic parameters compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria for subjects:

* Informed consent as documented by signature
* Confirmed biallelic mutation of cystathionine beta-synthase deficiency gene (homozygous or compound heterozygous) in an accredited Laboratory
* Continuation of their regular treatment under same dose (e.g. vitamin B6, B9 and B12, betaine) as prior to the study inclusion

Inclusion Criteria for controls:

- Healthy

Exclusion Criteria:

* Any clinically instable concomitant disease
* Individuals with acute cardiac events, syncope, rhythm disturbances or unstable hypertension in the past 6 months
* Individuals with vitamins B9 or B12 deficiencies
* Homocysteine > 100 µmol/l (for subjects)
* Homocysteine > 20 µmol/l (for controls)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Endocrinology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Plasma homocysteine concentration | -90 minutes before exercise to 24 hours after a 30 minute exercise
  Change in homocysteine concentration after a 30 minute exercise at fixed wattage

SECONDARY OUTCOMES:
Dietary parameters | During 3 days before and on the day of the exercise (day 1)
  self-reporting daily food diary
Indirect calorimetry | -90 minutes before exercise to the end of exercise (+30 minutes)
  Energy expenditure
Plasma amino acid profile | -90 minutes before exercise to 24hours after a 30 minute exercise
  Change in amino acid profile after a 30 minute exercise at fixed wattage
Plasma Insulin concentration | -90 minutes before exercise to 24 hours after a 30 minute exercise
  Change in insulin concentration after a 30 minute exercise at fixed wattage
Plasma lactate concentration | -90 minute before exercise to 24 hours after a 30 minute exercise
  Change in lactate concentration after a 30 minute exercise at fixed wattage
Plasma glucagon concentration | -90 minute before exercise to 24 hours after a 30 minute exercise
  Change in glucagon concentration after a 30 minute exercise at fixed wattage
Plasma free fatty acids concentration | -90 minute before exercise to 24 hours after a 30 minute exercise
  Change in free fatty acids concentration after a 30 minute exercise at fixed wattage
Plasma ketone bodies concentration | -90 minute before exercise to 24 hours after a 30 minute exercise
  Change in ketone bodies concentration after a 30 minute exercise at fixed wattage
Plasma cortisol concentration | -90 minute before exercise to 24 hours after a 30 minute exercise
  Change in cortisol concentration after a 30 minute exercise at fixed wattage
Blood pressure | -90 min before exercise to 24 hours after a 30 minute exercise
  Change in blood pressure after a 30 minute exercise at fixed wattage

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Département de physiologie, Lausanne, Canton of Vaud
  - Lausanne University Hospitals, Lausanne, Canton of Vaud

IPD SHARING:
Plan to Share IPD: No